CLINICAL TRIAL: NCT07037771
Title: Phase 3 Study to Evaluate the Efficacy and Safety of Zodasiran in Adolescent and Adult Subjects With Homozygous Familial Hypercholesterolemia (YOSEMITE)
Brief Title: A Phase 3 Study of Zodasiran in Adolescent and Adult Subjects With Homozygous Familial Hypercholesterolemia (YOSEMITE)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROANG3-3001
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — zodasiran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- zodasiran (Experimental): 5 doses of zodasiran by subcutaneous (sc) injection (randomized period). 4 or 5 doses of zodasiran by sc injection (optional open-label period).
  Interventions: Drug: zodasiran Injection
- Placebo (Placebo Comparator): Calculated volume to match active treatment by sc injection (randomized period).
  4 or 5 doses of zodasiran by sc injection (optional open-label period)
  Interventions: Drug: zodasiran Injection; Drug: Placebo

INTERVENTIONS:
Drug: zodasiran Injection — ARO-ANG3 Injection
  Other Names: ARO-ANG3
Drug: Placebo — sterile normal saline (0.9% NaCl)
  Arms: Placebo

SUMMARY:
This multicenter, randomized, placebo-controlled study will evaluate the efficacy and safety of zodasiran subcutaneous (SC) injection in subjects 12 years of age and older with genetically or clinically diagnosed Homozygous familial hypercholesterolemia (HoFH). After completion of the double blind (DB) treatment period subjects will be eligible to continue in the optional open-label extension (OLE) period of the study. All placebo subjects who opt to continue will transition to active drug during the OLE Period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12 years, non pregnant, non lactating, do not plan to become pregnant during the study
* Body weight ≥35 kg at Screening as patients could theoretically be <35 kg as the study continues.
* HoFH based on a supportive genetic test or a clinical diagnosis (total cholesterol >500 mg/dL[13 mmol/L] OR treated LDL-C concentration of ≥300 mg/dL [≥8 mmol/L] either accompanied by TGs <300 mg/dL [3.4 mmol/L] AND both parents with documented total cholesterol >250 mg/dL [6.5 mmol/L] OR cutaneous or tendinous xanthoma before 10 years of age)
* LDL-C ≥70 mg/dL (1.8 mmol/L)
* Hemoglobin A1c (HbA1c) ≤9.5%
* Total bilirubin <2xULN, unless in previously confirmed cases of Gilbert's syndrome
* Alanine aminotransferase or aspartate aminotransferase <3×ULN
* On standard of care, maximally tolerated lipid-lowering therapy

Exclusion Criteria:

* Use of a hepatocyte-targeted siRNA within 365 days before Day 1 (except inclisiran, which is permitted; administration of inclisiran and study drug must be separated by at least 4 weeks)
* Use of an antisense oligonucleotide molecule within 3 months before Day 1
* Use of evinacumab within 3 months before Day 1
* Non-response to evinacumab, defined as LDL-C reduction <15% from baseline after 2 doses
* Use of any other investigational agent or device within 30 days or 5 half-lives (whichever is longer) before Day 1
* Use of systemic corticosteroids (unless used as replacement therapy for pituitary/adrenal disease with a stable regimen)
* Estimated glomerular filtration rate <30 mL/min

NOTE: Additional Inclusion/exclusion criteria may apply per protocol

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2027-08-20 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline to Month 12 in Fasting Low Density Lipoprotein Cholesterol (LDL-C) (Randomized period) | Baseline, Month 12

SECONDARY OUTCOMES:
Percent Change from Baseline to Month 12 in Fasting Apolipoprotein B (ApoB) (Randomized Period) | Baseline, Month 12
Percent Change from Baseline to Month 12 in Fasting Non-High Density Lipoprotein Cholesterol (non-HDL-C) (Randomized Period) | Baseline, Month 12
Change from Baseline to Month 12 in Fasting LDL-C (Randomized Period) | Baseline, Month 12
Area Under the Plasma Concentration Versus the Time Curve (AUC) from Baseline to Month 12 for Fasting LDL-C (Randomized Period) | Baseline, Month 12
Percent Change from Baseline to Month 12 in Fasting Triglycerides (TGs) (Randomized Period) | Baseline, Month 12
Percent Change from Baseline to Month 12 in Fasting Angiopoietin-like Protein 3 (ANGPTL3) (Randomized Period) | Baseline, Month 12
Percent Change from Baseline to Month 12 in Fasting Total Cholesterol (Randomized Period) | Baseline, Month 12
Percent Change from Baseline to Month 12 in Fasting High-Density Lipoprotein Cholesterol (HDL-C) (Randomized Period) | Baseline, Month 12
Proportion of Participants who Meet European Union (EU) LDL-C Apheresis Eligibility Criteria (per German Apheresis Working Group) at Month 12 (Randomized Period) | Month 12
Proportion of Participants who Meet United States (US) Apheresis Eligibility Criteria (per National Lipid Association) at Month 12 (Randomized Period) | Month 12
Proportion of Participants with Fasting LDL-C <100 mg/dL (2.6 mmol/L) at Month 12 (Randomized Period) | Month 12
Change from Baseline in Fasting LDL-C Over Time (Randomized Period) | Baseline, Day 1, Months 1, 2, 3, 4.5, 6, 7.5, 9, 10.5, and 12
Percent Change from Baseline in fasting LDL-C Over Time (Randomized Period) | Baseline, Day 1, Months 1, 2, 3, 4.5, 6, 7.5, 9, 10.5, and 12
Percent Change from Baseline to Month 12 in Fasting Lipoprotein(a) [Lp(a)] (Randomized Period) | Baseline, Month 12

CONTACTS AND LOCATIONS:
Locations (8):
- United States (3):
  - Research Site 7, Park Ridge, Illinois
  - Research Site 2, New York, New York
  - Research Site 1, Cincinnati, Ohio
- Research Site 3, Nedlands, Western Australia, Australia
- Canada (3):
  - Research Site 5, Vancouver, British Columbia
  - Research Site 6, Chicoutimi, Quebec
  - Research Site 4, Québec, Quebec
- Research Site 8, Cape Town, South Africa